CLINICAL TRIAL: NCT01124682
Title: Image Guided Dose Escalated Adaptive Bladder Radiotherapy
Brief Title: 3-Dimensional Conformal Radiation Therapy in Treating Patients With Bladder Cancer Who Have Undergone Transurethral Resection of the Bladder
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000671670; ICR-IDEAL; EU-21035; CCR-3217; MREC-09/H0801/40
Record Dates: First submitted 2010-05-14; First posted 2010-05-17 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2011-02

CONDITIONS: Bladder Cancer
Keywords: adenocarcinoma of the bladder; squamous cell carcinoma of the bladder; transitional cell carcinoma of the bladder; recurrent bladder cancer; stage II bladder cancer; stage III bladder cancer; stage IV bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Radiotherapy, Conformal; Radiotherapy, Image-Guided; Serotonin Plasma Membrane Transport Proteins

INTERVENTIONS:
Procedure: diagnostic cystoscopy
Procedure: diffusion-weighted magnetic resonance imaging
Procedure: implanted fiducial-based imaging
Procedure: quality-of-life assessment
Radiation: 3-dimensional conformal radiation therapy
Radiation: image-guided radiation therapy
Radiation: selective external radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue.

PURPOSE: This phase I trial is studying the side effects and best dose of 3-dimensional conformal radiation therapy in treating patients with bladder cancer who have undergone transurethral resection of the bladder.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum-tolerated dose of external-beam radiotherapy delivered as a tumor boost in patients who have undergone prior transurethral bladder resection for muscle-invasive carcinoma of the bladder.

Secondary

* To document progression-free survival and overall survival of these patients.
* To evaluate patterns of recurrence and bladder preservation rates following dose-escalated radiotherapy in these patients.
* To determine the impact of acute and late toxicity on quality of life in these patients.
* To assess the use of gold seeds for tumor boost delineation in these patients.
* To evaluate the use of virtual cystoscopy tumor localization in these patients.
* To assess coverage of the phase II radiotherapy boost volume on the daily cone-beam images.
* To assess coverage of the phase III radiotherapy volume on cone-beam images with selected adaptive strategy.
* To evaluate the use of diffusion-weighted MRI (dwMRI) scans in assessing response to radiotherapy.

OUTLINE: This is a dose-escalation study.

Patients undergo a rigid cystoscopy and gold-seed insertion, if clinically appropriate. Approximately 3-5 seeds are inserted into the bladder wall to demarcate the maximum extent of visible tumor or tumor bed via a customized introducer. All patients undergo 3-dimensional conformal radiotherapy once daily, 5 days per week during weeks 1 and 4-7 and once daily, 4-6 days per week during weeks 2 and 3, using a combination of image-guided radiotherapy techniques and a partial bladder radiotherapy boost.

Patients complete quality-of-life questionnaire QOL-30 at baseline, 1 and 3 months, and then annually after completion of study treatment.

After completion of study treatment, patients are followed up at 4, 8, and 12 weeks, every 6 months for 3 years, and then annually for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive bladder carcinoma, including the following cellular types:

  * Adenocarcinoma
  * Transitional cell carcinoma
  * Squamous cell carcinoma
* Clinical stage G1-3, pT2a-4 disease

  * Localized disease
  * No bone or visceral metastases
  * No lymph node metastases
* Has undergone maximal transurethral resection of the bladder tumor and planning to receive radical radiotherapy

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Hemoglobin > 10 g/dL
* WBC > 3,000/mm^3
* Platelet count > 150,000/mm^3
* Creatinine < 120 μmol/L
* Bilirubin < 1.5 times upper limit normal (ULN)
* AST < 1.5 times ULN
* Alkaline phosphatase < 1.5 times ULN
* Not pregnant
* No inflammatory bowel disease or other significant small bowel disease
* Physically fit for radical radiotherapy
* No psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* No other malignancy within the past 2 years except adequately treated basal cell carcinoma of the skin or adequately treated carcinoma in situ of the cervix uteri

  * Prior superficial transitional cell carcinoma of the bladder allowed

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior pelvic surgery
* No bilateral hip replacements compromising accurate radiotherapy planning
* No prior radiotherapy to the pelvis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-05; Primary Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Maximum-tolerated dose

SECONDARY OUTCOMES:
Progression-free survival
Overall survival
Bladder preservation rates
Acute and late toxicity and safety profile
Quality of life
Tumor boost volumes delineated with and without gold seeds
Dose-volume histogram analysis of PTV2 and PTV3 coverage
Change in diffusion coefficient between pre- and post-radiotherapy dwMRI scans

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Huddart, MD, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden - Surrey, Sutton, England, United Kingdom